CLINICAL TRIAL: NCT01087008
Title: Assessment of the Antitumour Effect of Zoledronic Acid in Patients With Multiple Myeloma and Asymptomatic Biochemical Relapse: Prospective Clinical Trial of the GEM/PETHEMA Group
Brief Title: Zoledronic Acid in Patients With Multiple Myeloma and Asymptomatic Biochemical Relapse
Acronym: AZABACHE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Dynamic Solutions (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AZABACHE: 2009-017440-13
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Zoledronic acid
MeSH Terms: conditions — Multiple Myeloma | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronate acid (Experimental)
  Interventions: Drug: zoledronic acid
- No treatment control (Other)
  Interventions: Other: No treatment control

INTERVENTIONS:
Drug: zoledronic acid — Zoledronic acid 4 mg every 4 weeks for a total of 12 treatments
  Arms: Zoledronate acid
Other: No treatment control — Patients doesn't receive treatment
  Arms: No treatment control

SUMMARY:
Assessment of the antitumour effect of zoledronic acid in patients with multiple myeloma and asymptomatic biochemical relapse

It´s proposed to investigate the use of Zoledronic acid as single therapy in patients with Multiple Myeloma in biochemical relapse. The following must be noted:

* Patients with no formal indication for chemotherapy treatment will be included, as patients with symptomatic myeloma who after responding show biochemical relapse are generally not treated. This allows for generating both a group of patients untreated, on no additional treatment and a treatment group on zoledronic acid.
* As these are relapsing symptomatic patients, their number is far higher than patients with quiescent Multiple Myeloma. This allows for expecting a good enrolment.
* There are few reliable data on symptom progression after biochemical relapse, though it is one of the new objectives occurring in almost all clinical trials on myeloma. In the VISTA study, it has been estimated that the median time to the new treatment is 5 months (combining progression-free time and time to the next treatment). This time is much shorter than the median quiescent myeloma progression-free survival, so a very long follow-up time will not be necessary in this patient group.
* The administration of this drug to these patients can help prevent skeleton-related complications in the future, the study of which will be a secondary objective of this study.

DETAILED DESCRIPTION:
Zometa is administrated every 4 weeks at dose of 4 mg. The limit of administrations is 12. The first infusion is in the visit 2 and the last is in visit 13

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years.
* Signed informed consent before performing any study procedure that is not the part of the regular medical care of the patients.
* Diagnosis of MM, with biochemical relapse after initial response with no symptoms resulting from the disease (CRAB), defined as a re-positivation of a previous immunofixation (two samples) or increase above 25% of serum or urine protein M.
* In the investigator's opinion, ability to meet all clinical trial requirements

Exclusion Criteria:

* Treatment with bisphosphonates (oral route and/or endovenous route) within 3 months prior to inclusion.
* Treatment with denosumab within three months prior to inclusion.
* Criteria of symptomatic disease or organic damage related to disease, defined as:

  * Impaired renal function: serum creatinine >2 mg/dl or 173 mmol/l. Calcium increase: serum calcium ≥12 mg/dl within 28 days prior to inclusion.
* Anaemia: haemoglobin < 10 g/dl or 2 g/dl below normal ranges.
* Bone injury: new osteolytic lesions (from diagnosis) seen within 3 months prior to inclusion, current pathological fractures or increase of osteopenia (from diagnosis) in bone radiology series.
* Others: amyloidosis with current organic damage, recurrent bacterial infections (more than 2 events in 12 months), symptomatic hyperviscosity, presence of plasmacytomas.
* Patients with current and active dental disorders (dental, jaw infection, bone exposed in the mouth, jaw osteonecrosis).
* Patients developing jaw osteonecrosis or other serious adverse events due to treatment with any bisphosphonate .
* Significant liver disease:
* Bilirubin > 3 g/dl.
* ALT > 2.5 x the upper limit of normal
* AST > 2.5 x the upper limit of normal
* Patients who are currently in another clinical trial or receiving any investigational agent.
* Pregnancy or nursing.
* Parathyroid gland diseases.
* Previous malignancy with a high risk of death or bone disease: breast cancer, prostate cancer or lung cancer, even if on complete response.
* Active presence of neoplasms other than Multiple Myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2010-04 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-06-05 (Actual)

PRIMARY OUTCOMES:
Time to next need treatment | 6 months
  Time to the next treatment, considered as the time from the randomization date to the start of the next chemotherapy treatment for Multiple Mieloma or death for any cause

SECONDARY OUTCOMES:
Time to symptom relapse | 1 year
  Time to symptom relapse, considered as the time from randomization to symptom relapse
disease progression | 2 years
  To describe the differences between patients treated with ZOL or not in terms of type of disease progression (bone and extra-bone).
prognostic factors | 2 years
  To describe the prognostic factors in patients with MM and asymptomatic biochemical relapse
antitumour effect of ZOL | 1 year
  To assess the antitumour effect of ZOL on other clinically significant parameters in MM, including tumour response to ZOL
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: García Sanz Ramon, Dr, Study Chair — PETHEMA Foundation
Locations (16):
- Spain (16):
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Jose María Morales Meseguer, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Llàtzer, Palma de Mallorca
  - Hospital Universitario Son Dureta, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset., Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza

REFERENCES:
- [Result] R. García-Sanz, A. Oriol, J. de la Rubia, L. Palomera, P. Ribas, MT. Hernández, MJ. Moreno, J. Bargay, A. Ramírez, AI. Teruel, MJ. Blanchard, M. Gironella, M. Granell, E. Abellá, MA Sampol, R. Martínez, JF San Miguel EVALUTION OF BENEFITS AND POTENTIAL ANTIMYELOMA EFFECT OF ZOLEDRONIC ACID IN PATIENTS WITH ASYMPTOMATIC BIOCHEMICAL RELAPSES. Abstract for ASH 2012
- [Result] R. García-Sanz, A. Oriol, J. de la Rubia, L. Palomera, P. Ribas, MT. Hernández, MJ. Moreno, J. Bargay, A. Ramírez, AI. Teruel, MJ. Blanchard, M. Gironella, M. Granell, E. Abellá, MA Sampol, R. Martínez, JF San Miguel EVALUTION OF BENEFITS AND POTENTIAL ANTIMYELOMA EFFECT OF ZOLEDRONIC ACID IN PATIENTS WITH ASYMPTOMATIC BIOCHEMICAL RELAPSES. Abstract for EHA 2012
- [Result] R. García-Sanz, A. Oriol, J. de la Rubia, L. Palomera, P. Ribas, MT. Hernández, MJ. Moreno, J. Bargay, A. Ramírez, AI. Teruel, MJ. Blanchard, M. Gironella, M. Granell, E. Abellá, MA Sampol, R. Martínez, JF San Miguel EVALUTION OF BENEFITS AND POTENTIAL ANTIMYELOMA EFFECT OF ZOLEDRONIC ACID IN PATIENTS WITH ASYMPTOMATIC BIOCHEMICAL RELAPSES. Poster for EHA 2012
- [Derived] Garcia-Sanz R, Oriol A, Moreno MJ, de la Rubia J, Payer AR, Hernandez MT, Palomera L, Teruel AI, Blanchard MJ, Gironella M, Ribas P, Bargay J, Abella E, Granell M, Ocio EM, Ribera JM, San Miguel JF, Mateos MV; Spanish Myeloma Group (GEM/PETHEMA). Zoledronic acid as compared with observation in multiple myeloma patients at biochemical relapse: results of the randomized AZABACHE Spanish trial. Haematologica. 2015 Sep;100(9):1207-13. doi: 10.3324/haematol.2015.128439. Epub 2015 Jun 11. PMID 26069291
- See also: Novartis web page — http://www.novartis.es
- See also: Spnish Association of Haematology — http://aehh.org